CLINICAL TRIAL: NCT04040244
Title: A Pilot Study of Exhaled Breath Analysis to Predict Risk of Symptomatic Pneumonitis After Chemoradiotherapy For Stage III Non-Small Cell Lung Cancer
Brief Title: Exhaled Breath Analysis to Predict Risk of Symptomatic Pneumonitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI is requesting this study to be closed due to the departure of the Co-PI who is an integral part of the study.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00059924; WFBCCC 98119 (Other: Wake Forest Baptist Comprehensive Cancer Center); NCI-2019-05682 (Other: NCI); P30CA012197 (NIH)
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Results first posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-08

CONDITIONS: Pneumonitis; Nonsmall Cell Lung Cancer Stage III
MeSH Terms: conditions — Pneumonia; Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exhaled Breath Analysis (Experimental): Exhaled breathe condensate will be collected using R-tube and ReCIVA device over 5-10 minutes.
  Interventions: Other: Exhaled Breath Collection; Other: Blood sample

INTERVENTIONS:
Other: Exhaled Breath Collection — Exhaled breath condensate (EBC) and exhaled breath volatiles (EBV) samples will be obtained over 5-10 minutes using a one-time use R-tube apparatus.
Other: Blood sample — Blood samples collected simultaneously with routine standard of care blood draws.

SUMMARY:
This is a prospective pilot study investigating exhaled breath condensate analyses to quantify the variability over time of various biomarkers associated with symptomatic pneumonitis.

DETAILED DESCRIPTION:
Primary Objective:

• To quantify the intra-person variability of concentrations of TGF-β1, IL-6, IL-1α, and IL-10 measured in exhaled breath condensate.

Secondary Objectives:

* To examine the associations between differences in pre-treatment and post-treatment exhaled breath condensate concentrations of TGF-β1, IL-6, IL-1α, and IL-10 and the development of CTCAE grade 2+ symptomatic pneumonitis.
* To examine the associations between serum measures of TGF-β1, IL-6, IL-1α, and IL-10 and:
* Exhaled breath condensate measures of the same biomarkers, and
* The development of CTCAE grade 2+ symptomatic pneumonitis.
* To examine the association between microbiome signatures found in pre-treatment exhaled breath condensate and the development of CTCAE grade 2+ symptomatic pneumonitis.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old.
* Clinically diagnosed or suspected Stage III non-small cell lung cancer to be treated with chemoradiotherapy as part of cancer treatment, as determined by the treating clinician.
* Plan for treatment with definitive radiotherapy (≥60 Gy) with concurrent chemotherapy at the discretion of the treating radiation and medical oncologists.
* Willing and able to tolerate exhaled breath collection.
* Able to provide informed consent.

Exclusion Criteria:

* Systemic (oral, intravenous or intramuscular) corticosteroid use for any reason within 5 days of registration.
* Prior radiotherapy directed at the chest (thoracic inlet superiorly to diaphragm inferiorly).
* Any systemic antibiotic use within 2 weeks of registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Farris, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exhaled Breath Analysis
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exhaled Breath Analysis
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 65.6 [53 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Variability of Biomarkers
Description: Concentrations of TGF-β1, IL-6, IL-1α, and IL-10 (ng/mL) will be measured in exhaled breath condensate at baseline, at 2 weeks and after chemotherapy start and 6 weeks after chemotherapy start (the end of chemotherapy) and 1 month after completion of chemotherapy using a 2-tailed alpha of 0.05 with detectable standard deviation units from baseline to post treatment.
Time Frame: At baseline and one month after completion of chemotherapy
Population: 9 have data at baseline; 6 have data at 1 month post CRT (chemo-radiation treatment)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Exhaled Breath Analysis
Number analyzed (Participants) | 9
ng/mL
  TGF-b1 baseline | 87.84 (15.94)
  TGF-b1 1 month post CRT: number analyzed (Participants) | 6
  TGF-b1 1 month post CRT | 100.47 (21.90)
  IL-6 baseline | 5.39 (2.49)
  IL-6 1 month post CRT: number analyzed (Participants) | 6
  IL-6 1 month post CRT | 6.96 (1.11)
  IL-10 baseline | 136.91 (19.85)
  IL-10 1 month post CRT: number analyzed (Participants) | 6
  IL-10 1 month post CRT | 151.07 (26.99)
  IL-1a baseline | 2.41 (2.52)
  IL-1a 1 month post CRT: number analyzed (Participants) | 6
  IL-1a 1 month post CRT | 2.36 (9.72)

2. Secondary Outcome: Differences in Concentrations of Biomarkers in Exhaled Breath Condensate From Baseline to 1 Month Post CRT
Description: TGF-β1, IL-6, IL-1α, and IL-10 (ng/mL) measured in exhaled breath condensate to compare mean change levels from (baseline), at 2 weeks after CRT start, 6-weeks after CRT start (the end of CRT), and 1 month after completion of chemotherapy using t-tests comparing mean change levels in each marker.
Time Frame: One month after completion of chemotherapy
Population: 6 participants who had relevant data at both required time points
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Exhaled Breath Analysis
Number analyzed (Participants) | 6
ng/mL
  TGF-b1 mean diff | 14.81 (18.17)
  IL-6 mean diff | 1.03 (2.34)
  IL-10 mean diff | 18.62 (24.15)
  IL-1a mean diff | 2.36 (9.72)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Exhaled Breath Analysis
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 5/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exhaled Breath Analysis (N=16)
Hypotension (Vascular disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Gastrointestional hemorrhage (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exhaled Breath Analysis (N=16)
Cardiac disorders (Cardiac disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) — Heartburn
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pharyngitis (Infections and infestations) | 1 (1)
Noncardiac chest pain (General disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT04040244/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT04040244/ICF_000.pdf